CLINICAL TRIAL: NCT00421122
Title: A 6-Month, Phase IIIA, Multi-Center,Randomised,Double-Blind, Double-Dummy, Parallel-Group Study of the Efficacy and Safety of Symbicort® Turbuhaler®+ Bricasol® pMDI Compared With Pulmicort® Turbuhaler®+Bricasol® pMDI in Chinese Patients With COPD
Brief Title: Efficacy and Safety Study of Symbicort Turbuhaler in Chinese Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D5892C00013
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chinese patients; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination; Terbutaline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 1 (Active Comparator): Bricasol®
  Interventions: Drug: terbutaline sulfate (Bricasol)
- 2 (Experimental): Bricasol® + Pulmicort®
  Interventions: Drug: budesonide (Pulmicort); Drug: terbutaline sulfate (Bricasol)
- 3 (Experimental): Bricasol® + Symbicort®
  Interventions: Drug: budesonide/formoterol (Symbicort); Drug: terbutaline sulfate (Bricasol)

INTERVENTIONS:
Drug: budesonide/formoterol (Symbicort) — inhalation therapy
  Other Names: Symbicort® Turbuhaler
  Arms: 3
Drug: budesonide (Pulmicort) — inhalation
  Other Names: Pulmicort® Turbuhaler
  Arms: 2
Drug: terbutaline sulfate (Bricasol) — inhalation therapy
  Other Names: Bricasol pMDI

SUMMARY:
This study aims at evaluating efficacy and safety of Symbicort® Turbuhaler® in Chinese COPD patients as defined by GOLD treatment guidelines in order to obtain an approval for indication of COPD from Chinese State Food and Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated inform consent
* Out-patient, clinical diagnosis of COPD
* Men or women at the age of 40 or over

Exclusion Criteria:

* A history of asthma
* Seasonal allergic rhinitis before 40 years of age
* Patients with significant or unstable ischemic heart disease, arrhythmia, cardiomyopathy, heart failure, uncontrolled hypertension as defined by the investigator or other disorder

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2006-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Post-study medication FEV1 | 1 hour after medication

SECONDARY OUTCOMES:
FVC | Pre dose and 1 hour post dose
FEV1 | Pre-dose and 15 minutes post dose
SGRQ symptom scores
COPD symptom scores
morning and evening PEF | Assessed daily
reliever medication use
AE
lab measures
ECG
physician examination
vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Symbicort Medical Science Director, MD, Study Director — AstraZeneca
Locations (8):
- China (8):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Nanjing, Jiangsu
  - Research Site, Shenyang, Liaoling
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Xi’an, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Hangzhou, Zhejiang

REFERENCES:
- [Derived] Zhong N, Zheng J, Wen F, Yang L, Chen P, Xiu Q, Yao W, Sun T, Zhao Z, Shen H, Shi Y, Lin J, Li Q. Efficacy and safety of budesonide/formoterol via a dry powder inhaler in Chinese patients with chronic obstructive pulmonary disease. Curr Med Res Opin. 2012 Feb;28(2):257-65. doi: 10.1185/03007995.2011.636420. Epub 2012 Jan 20. PMID 22046961